CLINICAL TRIAL: NCT02876237
Title: Patient Over 75 Years With Prostate Cancer: Geriatric Determinants of General Repercussion of Radiotherapy With Curative Intent
Brief Title: Geriatric Determinants of General Repercussion of Radiotherapy for Patient Over 75 Years With Prostate Cancer
Acronym: PROGERAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICO-A-2014-04; 2014-A00300-47 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2016-07-22; First posted 2016-08-23 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Geriatric Assessment; Quality of Life; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- geriatric assessment and quality of life (Experimental): Included patient must have a geriatric assessment before radiotherapy and 6 months later.
  Patient must complete quality of life questionnaire before radiotherapy then 2 and 6 months later.
  Interventions: Other: geriatric assessment and quality of life; Radiation: Radiotherapy

INTERVENTIONS:
Other: geriatric assessment and quality of life — Included patient must have a geriatric assessment before radiotherapy and 6 months later. This standardized geriatric assessment will collect social information, functional, sensory, cognitive, emotional, motor, nutritional, and medical related to comorbidities .
  Patient must complete quality of life questionnaire before radiotherapy then 2 and 6 months later.
Radiation: Radiotherapy — standard radiotherapy

SUMMARY:
The investigators propose to carry out a prospective analysis of physical impact, psychological, cognitive and social of radiotherapy in all patients over 75 years bearer of localized prostate cancer with an indication of curative radiotherapy. This standardized geriatric assessment will collect social information, functional, sensory, cognitive, emotional, motor, nutritional, and medical related to comorbidities . The quality of life of patients will be evaluated by the QLQ C30 (Quality of Life Questionnaire) European Organisation for Research and Treatment of Cancer (EORTC) before starting treatment, at the end of radiotherapy (2 months) and at 6 months. This short follow-up period seems appropriate in this elderly population and will allow an answer within 2 years to the problem raised in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Man with a histologically proven prostate cancer
2. Indication of a curative intent radiotherapy
3. Age ≥ 75 years
4. Patient who signed an informed consent

Exclusion Criteria:

1. Patient with metastatic prostate cancer
2. Patient unable to submit to monitoring of the protocol for social, geographical or family reasons
3. A person who is not affiliated to a social security scheme or of such a scheme
4. Patient under trusteeship

Min Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 230 (Actual)
Dates: Start 2015-02; Primary Completion 2017-02 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
General tolerance of the radiotherapy evaluated by the QLQ-C30 questionnaire | 2 months
  Tolerance will be called bad for the loss of 20 or more points (out of 100) between the initial assessment and evaluations at 2 and 6 months. Tolerance will be called correct in other cases. This threshold of 20 points was selected according to the work of Osoba.
Complete geriatric assessment | 6 months
  This standardized geriatric assessment will collect social information, functional, sensory, cognitive, emotional, motor, nutritional, and medical related to comorbidities .
General tolerance of the radiotherapy evaluated by the QLQ-C30 questionnaire | 6 months
  Tolerance will be called bad for the loss of 20 or more points (out of 100) between the initial assessment and evaluations at 2 and 6 months. Tolerance will be called correct in other cases. This threshold of 20 points was selected according to the work of Osoba.

CONTACTS AND LOCATIONS:
Overall Officials: Aurore GOINEAU, MD, Principal Investigator — Institut de Cancerologie de l'Ouest; Stéphane SUPIOT, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (10):
- France (10):
  - Institut de Cancérologie de l'Ouest, Angers
  - Hopital Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - CHD, La Roche-sur-Yon
  - Centre Hospitalier Bretagne Sud, Lorient
  - Centre Catherine de Sienne, Nantes
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - CHP, Saint-Grégoire
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Institut de Cancérologie de Loire, Saint-Priest-en-Jarez